CLINICAL TRIAL: NCT00002044
Title: A Pilot Study To Evaluate the Effect of Retrovir (Zidovudine: AZT) in the Treatment of Human Immunodeficiency Virus (HIV) Associated Dementia and Neuromuscular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 014D; 14
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-02

CONDITIONS: AIDS Dementia Complex; Neuromuscular Diseases; HIV Infections
Keywords: Pilot Projects; Neuromuscular Diseases; Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS Dementia Complex; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — AIDS Dementia Complex; Neuromuscular Diseases; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
The purpose of this pilot study is to evaluate the efficacy of Retrovir (AZT) in the treatment of AIDS-related dementia and various neuromuscular complications. HIV is both a lymphotropic and neurotropic virus which can affect both the central and peripheral nervous systems (CNS, PNS). There is evidence that the CNS and PNS may harbor the virus in a latent state, with the potential for continuous reinfection of other body systems. Therefore, effective therapeutic efforts against HIV infection should provide effective antiviral activity within the nervous system.

ELIGIBILITY:
Inclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Past or present renal disease.
* Significant bone marrow suppression.
* Blood transfusion within the past month.
* Liver dysfunction.
* Evidence of an underlying, severe infection.
* Evidence of an active life-threatening opportunistic infection at study entry.
* Severe malabsorption (patients with recent significant weight loss must have a serum carotene level of > 75 IU/ml).
* Evidence of nervous system dysfunction being caused by factors other than HIV infection, particularly by cerebral toxoplasmosis, lymphoma, cryptococcal meningitis, chronic alcohol abuse, lead poisoning, cytomegalovirus (CMV) infection (patients with retinal CMV infection or other evidence of CMV dementia), syphilis, or progressive multifocal leukoencephalopathy.
* Other known causes of nerve or muscle disease.
* Hypersensitivity to zidovudine (AZT).
* Lymphoma or other tumor requiring cytotoxic chemotherapy.

Concurrent Treatment:

Allowed:

* Electron beam therapy to an area of less than 100 cm2.

Patients with the following are excluded:

* Past or present renal disease.
* Significant bone marrow suppression.
* Blood transfusion within the past month.
* Liver dysfunction.
* Evidence of an underlying, severe infection.
* Evidence of an active life-threatening opportunistic infection at study entry.
* Severe malabsorption (patients with recent significant weight loss must have a serum carotene level of > 75 IU/ml).
* Evidence of nervous system dysfunction being caused by factors other than HIV infection, particularly by cerebral toxoplasmosis, lymphoma, cryptococcal meningitis, chronic alcohol abuse, lead poisoning, cytomegalovirus (CMV) infection (patients with retinal CMV infection or other evidence of CMV dementia), syphilis, or progressive multifocal leukoencephalopathy.
* Other known causes of nerve or muscle disease.
* Hypersensitivity to zidovudine (AZT).
* Lymphoma or other tumor requiring cytotoxic chemotherapy.

Patients with AIDS (CDC surveillance definition) or AIDS related complex (ARC).

* All patients must have either:
* Dementia as defined by a progressive cognitive impairment in the absence of altered consciousness that is thought to be causally related to HIV infection. Patients in this study will fall into the lower 20 percent (or less) of a normal sample of formal neuropsychological testing.
* OR
* One of the following neuromuscular diseases thought to be related to HIV infection:
* Demyelinating polyneuropathy, axonal polyneuropathy, inflammatory myopathy, or unexplained progressive muscle weakness.
* Capacity to give informed consent or a person with durable power of attorney who can give informed consent.
* Life expectancy = or > 4 months.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Cytotoxic chemotherapy.
* Steroids.
* Interferon.
* Immunomodulating agents.

Concurrent Treatment:

Excluded:

* Radiation therapy (except electron beam therapy to an area of less than 100 cm2).

Prior Medication:

Excluded within 4 weeks of study entry:

* Cytotoxic chemotherapy.
* Any retroviral drug including but not limited to zidovudine (AZT), ribavirin, HPA 23, AL721, or phosphonoformate.
* Steroids.
* Interferon.
* Immunomodulating agents.
* An anticipated need for any of these agents within the next 16 weeks.

Prior Treatment:

Excluded within 1 month of study entry:

* Radiation therapy (except electron beam therapy to an area of less than 100 cm2).
* Blood transfusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States